CLINICAL TRIAL: NCT04523506
Title: The Effects of Botulinum Toxin on Oral Aperture in Patients With Scleroderma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Heather Woodworth Goff, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0169
Record Dates: First submitted 2020-07-19; First posted 2020-08-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- the temporomandibular joint (TMJ) group (Experimental): This study will evaluate the use of botulinum toxin for microstomia (reduced oral aperture) in scleroderma patients. The TMJ group will be injected with two units of Botox into four different injection points to each masseter (16 units of Botox total) at the initial visit. No additional Botox will be injected in subsequent visits. Botox is a neurotoxin that functions as a paralytic by preventing the release of acetylcholine to inhibit muscle contracture and decrease fibrosis by decreasing differentiation of fibroblasts to myofibroblasts, decreasing expression of collagen, and increasing expression of matrix metalloproteinase1
  Interventions: Biological: Botulinum toxin(Botox)
- the perioral group (Experimental): Biological/Vaccine: Botulinum toxin(Botox) This study will evaluate the use of botulinum toxin for microstomia (reduced oral aperture) in scleroderma patients. The perioral group will be injected with two units of Botox into eight different injection points (16 units of Botox total) around the lips (in the orbicularis oris). Botox is a neurotoxin that functions as a paralytic by preventing the release of acetylcholine to inhibit muscle contracture and decrease fibrosis by decreasing differentiation of fibroblasts to myofibroblasts, decreasing expression of collagen, and increasing expression of matrix metalloproteinase1-3.
  Interventions: Biological: Botulinum toxin(Botox)

INTERVENTIONS:
Biological: Botulinum toxin(Botox) — This study will evaluate the use of botulinum toxin for reduced oral aperture in scleroderma patients. Botox is a neurotoxin that functions as a paralytic by preventing the release of acetylcholine to inhibit muscle contracture and decrease fibrosis by decreasing differentiation of fibroblasts to myofibroblasts, decreasing expression of collagen, and increasing expression of matrix metalloproteinase.

SUMMARY:
This study will evaluate the use of botulinum toxin for microstomia (also known as reduced oral aperture) in scleroderma patients. Botox is a neurotoxin that functions as a paralytic by preventing the release of acetylcholine to inhibit muscle contracture and decrease fibrosis by decreasing differentiation of fibroblasts to myofibroblasts, decreasing expression of collagen, and increasing expression of matrix metalloproteinase1-3. The study will include three arms: the temporomandibular joint (TMJ) group who will receive injections of Botox to the masseter, the perioral group who will receive injections of Botox around the lips, and a control group who will receive no treatment for ROA. Outcome measurements will include measurement of oral aperture size through measurement inter-labial distance and between the upper and lower lips and the inter-incisal distance, patient satisfaction via a Skindex16 survey, mouth disability via the Mouth Handicap in Systemic Sclerosis Scale (MHISS), and patient and physician satisfaction using the Visual Analogic Scale (VAS). The maximum number of subjects to be consented for this study is 30. The study is expected to last four months per subject from time of consent to last clinical evaluation. Conditions that may result in a subject exiting the study prior to completion date include non-compliance, withdrawal of consent, or safety concerns such as adverse events as a result of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ddiagnosis of scleroderma (defined by the 2013 Classification Criteria for Systemic Sclerosis4,5)23,24 ) who also have microstomia (reduced oral aperture), defined as an inter-incisal distance less than 50 mm 6-7)m13,14 .
2. Male and female subjects.
3. English and non-English speakers.
4. Subjects aged 18 years old to 65 years old will be considered

Exclusion Criteria

1. Patients under 18 years old will be excluded.
2. Patients with a known history of a hypersensitivity to any Botox formulation or to any of the components in the formulation,
3. Active skin infection at the proposed injection site.
4. Concomitant neuromuscular disorder.
5. Pregnant or lactating.
6. Missing incisors.
7. treatment with: cyclophosphamide, Ultraviolet A-1 therapy, or topical calcitriol..

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Changes in inter-labial distance | This will be measured at baseline before treatment, 2 weeks after treatment, and 3 months after treatment.
  Inter-labial distance is defined as the distance between the upper and lower lip at maximum mouth opening. Distance will be measured using digital calipers by the same operator
Changes interincisal distance | This will be measured at baseline before treatment, 2 weeks after treatment, and 3 months after treatment.
  Interincisal distance is defined by the didistance between upper and lower incisor at maximum mouth opening. Distance will be measured using digital calipers by the same operator
quality of life via a Skindex16 survey | This information will be collected at baseline before treatment, 2 weeks after treatment, and 3 months after treatment.
  This is a patient quality of life survey using the skindex 16 survey form.

SECONDARY OUTCOMES:
Changes in the inter-commissural distance | This will be measured at baseline before treatment, 2 weeks after treatment, and 3 months after treatment.]
  Inter-commissural distance is defined by the distance from corner to corner at the angle of the lip (also known as the oral commissures). Distance will be measured using digital calipers by the same operator.
Changes in the Mouth Handicap in Systemic Sclerosis Scale (MHISS) | This will be measured at baseline before treatment, 2 weeks after treatment, and 3 months after treatment.]
  Mouth disability will be assessed via the Mouth Handicap in Systemic Sclerosis Scale (MHISS). MHISS range from 0 to 48 with 48 being worse disability

CONTACTS AND LOCATIONS:
Overall Officials: Heather Goff, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas - Dermatology Clinical Trials, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be decided by research team